CLINICAL TRIAL: NCT04163705
Title: Immune Profile of Patients With Positive Blood Cultures and Multiple Organ Dysfunctions
Brief Title: Immune Profile of Patients With Sepsis
Acronym: IPSEPSIS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Nestor Pistillo, Head of Intensive Care Unit at Hospital El Cruce, Hospital El Cruce
Other Study IDs: Hospital El Cruce
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Sepsis, Severe
Keywords: Multiple organ dysfunctions
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — The plasma will be stored at -80 ° for later analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gram negative: The presence of one or more positive samples will be considered positive blood cultures.
  Patients with severe sepsis will be enrolled prospectively and consecutively. Some of the blood used for blood culture samples will be processed for the study (sample 0). The plasma will be stored at -80 ° for later analysis. A routine clinical and laboratory database will be completed.
  Only patients who have positive blood cultures will be randomized according to their result in: sepsis by Gram positive or Gram negative.
  Interventions: Diagnostic Test: blood sample collection
- Gram positive: The presence of one or more positive samples will be considered positive blood cultures.
  Patients with severe sepsis will be enrolled prospectively and consecutively. Some of the blood used for blood culture samples will be processed for the study (sample 0). The plasma will be stored at -80 ° for later analysis. A routine clinical and laboratory database will be completed.
  Only patients who have positive blood cultures will be randomized according to their result in: sepsis by Gram positive or Gram negative.
  Interventions: Diagnostic Test: blood sample collection

INTERVENTIONS:
Diagnostic Test: blood sample collection — Routine Laboratory Analysis

SUMMARY:
The immune response can acquire different profiles (proinflammatory and anti-inflammatory response) depending on the activating agent.The objective of this study is to compare the immunological profile in patients with severe sepsis and positive blood cultures.

DETAILED DESCRIPTION:
Sepsis is one of the leading causes of death in patients admitted to intensive care. It is characterized by being an exaggerated and deregulated inflammatory response triggered by an infection. Although inflammation affects the compartmentalization of the infection, the activation of the immune system in sepsis has a systemic problem, which sometimes affects the organs distant from the site of infection. Within this context, two processes are recognized, which can often coexist: the pro-inflammatory response and the anti-inflammatory response. While it is assumed that the proinflammatory response may favor the development of multiple organ failure, sepsis-induced immunosuppression would favor a new infection, especially of endogenous and intranosocomial germs, mortality increases. The pro-anti-inflammatory nature of sepsis (if so can be defined) depends on a multitude of factors: the type of infection, personal history, genetic conditions, associated diseases, environmental factors, the use of immunosuppressive medications and nutrition. state, among others. Recent studies found that the immune response profile differs depending on the type of infection (Gram negative or Gram positive). Defining the predominant immune condition is not a simple task. Here there are no commonly used clinical variables that define the immune status, except for neutrophil counts.

Objetive:

* Define whether there are differences in the immunological profile between patients with sepsis and positive blood cultures by Gram negative and Gram positive.
* Identify easily accessible clinical and / or laboratory patterns that can predict the predominant immune character.

Design: The study was approved by the Scientific and Ethics committee of the institution. Informed consent will be requested.

Patients with severe sepsis and positive blood cultures will be included prospectively, within 24 hours of diagnosis of sepsis.

Consider severe sepsis to life-threatening organic dysfunction caused by a deregulated host response to infection. This concept includes at least a score of the SOFA (sequential evaluation of organic insufficiency) scale equal to or greater than 2 points The presence of one or more positive samples will be considered positive blood cultures.

Patients with severe sepsis will be enrolled prospectively and consecutively. Some of the blood used for blood culture samples will be processed for the study (sample 0). The plasma will be stored at -80 ° for later analysis. A routine clinical and laboratory database will be completed.

Only patients who have positive blood cultures will be randomized according to their result in: sepsis by Gram positive or Gram negative.

Patients with severe sepsis but with negative blood cultures will be considered a control group. In patients with positive blood cultures, new blood samples will be taken between days 3 to 5 of sample 0 to define the evolution of the pro and anti-inflammatory response.

Minimum 12 patients per group will be included. The level of proinflammatory cytokines (TNF alpha and IL 1) and anti-inflammatory (IL10 and IL1 receptor) will be measured by ELISA method. Finally, the data will be analyzed and the differences between patients with Gram-positive and Gram-negative infections will be established.

Primary Outcome Measure:

Measurement of the pro-inflammatory and anti-inflammatory response in patients with severe sepsis and positive blood cultures

ELIGIBILITY:
Inclusion Criteria: severe sepsis -

Exclusion Criteria:

VIH immunosuppression Autoimmune disease Neoplasm Pregnant women Cirrhosis Bone Marrow Disease Malnutrition.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe sepsis and positive blood cultures will be included prospectively, within 24 hours of diagnosis of sepsis.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proinflammatory response. | Six months
  Plasma level comparison of: TNF-alpha, IL-6 and IL-1 between both groups, by flow cytometry.
Comparison of the anti-inflammatory response | Six months
  Plasma level comparison of: TNF-alpha receptor, INF-gamma and IL-10 between both groups, by flow cytometry.

SECONDARY OUTCOMES:
Mortality comparison | Six months
  Mortality between both groups will be compared for the 28th day of admission to the protocol.
SOFA score comparison | Six months
  Multiple organ dysfunction will be measured with the SOFA score at the time of admission to the protocol and between days 3 to 5. The severity score will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Pistillo, MD, Principal Investigator — Hospital El Cruce

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Gotts JE, Matthay MA. Sepsis: pathophysiology and clinical management. BMJ. 2016 May 23;353:i1585. doi: 10.1136/bmj.i1585. PMID 27217054
- [Background] Faix JD. Biomarkers of sepsis. Crit Rev Clin Lab Sci. 2013 Jan-Feb;50(1):23-36. doi: 10.3109/10408363.2013.764490. PMID 23480440
- [Background] Zeni F, Vindimian M, Pain P, Gery P, Tardy B, Bertrand JC. Antiinflammatory and proinflammatory cytokines in patients with severe sepsis. J Infect Dis. 1995 Oct;172(4):1171-2. doi: 10.1093/infdis/172.4.1171. No abstract available. PMID 7561209
- [Background] Endo S, Inada K, Inoue Y, Kuwata Y, Suzuki M, Yamashita H, Hoshi S, Yoshida M. Two types of septic shock classified by the plasma levels of cytokines and endotoxin. Circ Shock. 1992 Dec;38(4):264-74. PMID 1292890
- [Background] Annane D, Bellissant E, Cavaillon JM. Septic shock. Lancet. 2005 Jan 1-7;365(9453):63-78. doi: 10.1016/S0140-6736(04)17667-8. PMID 15639681
- [Background] Minasyan H. Sepsis and septic shock: Pathogenesis and treatment perspectives. J Crit Care. 2017 Aug;40:229-242. doi: 10.1016/j.jcrc.2017.04.015. Epub 2017 Apr 18. PMID 28448952
- [Background] Guenter CA, Hinshaw LB. Comparison of septic shock due to gram-negative and gram-positive organisms. Proc Soc Exp Biol Med. 1970 Jul;134(3):780-3. doi: 10.3181/00379727-134-34882. No abstract available. PMID 4988179
- [Result] Janols H, Bergenfelz C, Allaoui R, Larsson AM, Ryden L, Bjornsson S, Janciauskiene S, Wullt M, Bredberg A, Leandersson K. A high frequency of MDSCs in sepsis patients, with the granulocytic subtype dominating in gram-positive cases. J Leukoc Biol. 2014 Nov;96(5):685-93. doi: 10.1189/jlb.5HI0214-074R. Epub 2014 Jun 13. PMID 24929004